CLINICAL TRIAL: NCT05408260
Title: Feasibility of Automated Breast Ultrasound (ABUS) Versus Handheld Ultrasound (HHUS) for Breast Cancer Surveillance in Women With Nipple Sparing or Skin Sparing Mastectomy With Reconstruction
Brief Title: A Study to Compare the Effectiveness of Two Types of Ultrasound Technologies in Women Who Have Had Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 19D.799; JT 14405 (Other: JeffTrial Number)
Record Dates: First submitted 2022-06-02; First posted 2022-06-07 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Malignant Breast Neoplasm
MeSH Terms: conditions — Breast Neoplasms | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Screening (automated breast ultrasound, handheld ultrasound) (Experimental): Participants undergo HHUS and ABUS in no required order over 1 hour.
  Interventions: Procedure: Ultrasonography; Procedure: Automated Breast Ultrasound

INTERVENTIONS:
Procedure: Ultrasonography — Undergo HHUS
Procedure: Automated Breast Ultrasound — Undergo ABUS
  Other Names: ABUS

SUMMARY:
This clinical trial evaluates automated breast ultrasound (ABUS) and handheld ultrasound (HHUS) for the screening of women who have undergone breast reconstruction after breast cancer. Ultrasounds use high-frequency sound waves to create pictures of internal organs and tissues. ABUS has been found to be equal to HHUS for whole breast screening, but no data exist on its use for screening of reconstructed patients. This clinical trial evaluates the feasibility of using ABUS versus HHUS to screen women who have undergone reconstruction.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To show that ABUS reduces artifact compared to HHUS in terms of detection of the residual tissue in reconstructed nipple sparing mastectomy (NSM) and skin sparing mastectomy (SSM) patients.

SECONDARY OBJECTIVES:

I. To evaluate both the performance and interpretation times for ABUS and HHUS so that these factors can be considered when scheduling patients and for ease of implementation into practice.

II. A short survey will be administered immediately after both ultrasounds performed to enrolled patients to assess their experience with HHUS and ABUS, specifically addressing their perceived comfort level on a numerical scale and if they would be interested in obtaining subsequent annual screening HHUS or ABUS.

EXPLORATORY OBJECTIVE:

I. The appearance of native and reconstructed anatomy on ABUS and HHUS will be studied.

OUTLINE:

Participants undergo HHUS and ABUS in no required order over 1 hour.

Participants with ultrasound results indicating Breast Imaging Reporting and Data System (BI-RADS) 4 or 5 (suspicious and needs biopsy) undergo biopsy within 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Female
* >= 18 years of age at time of consent
* Free of focal breast symptoms and with no suspicious breast physical exam findings
* Previous unilateral NSM or SSM with implant (silicone, saline) or flap reconstruction performed at Thomas Jefferson University Hospital
* Must be able to understand and provide signed and dated informed consent form. If a patient understands the informed consent but is unable to sign, a legally authorized representative (LAR) may sign
* Willing to comply with all study procedures and be available for the duration of the study
* Willing to honor any bills that may be incurred if the insurance company does not pay for the billed bilateral hand held ultrasound

Exclusion Criteria:

* History of breast cancer recurrence
* Current focal breast symptoms since NSM or SSM with reconstruction
* NSM or SSM with reconstruction was performed years prior to study enrollment
* Bilateral NSM or SSM with reconstruction
* Females who are pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-11-18 (Actual); Primary Completion 2025-02-17 (Actual); Study Completion 2025-02-17 (Actual)

PRIMARY OUTCOMES:
Detection of the residual tissue (i.e., artifact) in reconstructed nipple sparing mastectomy (NSM) and skin sparing mastectomy (SSM) patients by automated breast ultrasound (ABUS) and handheld ultrasound (HHUS) | Up to 1 year
  This is a binary endpoint. The rate of artifact will be compared between handheld and automated scanning using McNemar test.

CONTACTS AND LOCATIONS:
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States